CLINICAL TRIAL: NCT00669851
Title: A Phase 3, International, Exploratory, Open-Label, Multicenter, Dual-Injection, Echocardiographic Imaging Settings and Safety Study of AI-700 in Normal Volunteers and Stable Cardiac Patients
Brief Title: Acquiring Consensus for Contrast Echocardiography System Settings - ACCESS Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Acusphere (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AI-700-34
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; echocardiography; cardiac imaging; heart disease; ultrasound contrast agent; myocardial contrast enhancement; myocardial perfusion
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases | interventions — perfluorobutane

INTERVENTIONS:
Drug: AI-700

SUMMARY:
This study evaluated and optimized settings for, and evaluated the performance of, AI-700-enhanced echocardiographic imaging on several ultrasound imaging platforms, as well as collected additional safety data for AI-700 in healthy volunteers and stable cardiac patients.

DETAILED DESCRIPTION:
Because the quality of AI-700-enhanced images is in part determined by the ultrasound (US) settings selection, the continuing study of different imaging modes and/or techniques is required in order to provide US settings recommendations for the many available systems. Therefore AI-700-enhanced imaging was performed in this study using imaging platforms and modes not previously tested and the AI-700 dose and administration methods employed in previous Phase 3 studies.

Two cohorts of subjects were studied at each site. Enrollment commenced with Cohort A and included normal (healthy) volunteers and stable cardiac patients. Settings optimization was performed in Cohort A using a single platform and real-time imaging. If the Sponsor agreed that the images and settings acquired in Cohort A were acceptable, the site was authorized to begin enrollment in Cohort B using the platform and settings that were defined in Cohort A. Authorized sites enrolled stable cardiac patients in Cohort B; no healthy volunteers were studied. For Cohort B subjects, the first 0.04 mL/kg dose of AI 700 was used to evaluate real-time imaging with the settings defined in Cohort A. The second dose of AI-700 for Cohort B subjects may have been used to confirm the data obtained with the first dose, or to explore imaging in a second mode (e.g. 3D/4D) and/or using real-time, high mechanical index triggered imaging on a second platform.

ELIGIBILITY:
Inclusion Criteria:

* For Cohort A, men and non-pregnant/non-lactating women in good health who are 18 to 70 years of age and who have a low chance of CAD will be enrolled.
* For Cohort B, men and non-pregnant/non-lactating women in good health who are 18-70 years of age who have had a prior MI and/or coronary artery revascularization intervention >90 days before AI-700 administration, without new or recurrent angina will be enrolled.

Exclusion Criteria:

* Healthy volunteers in Cohort A who have or have had any of the following conditions will be excluded from the study: clinically significant intra-cardiac shunts or any other cardiovascular structural and/or severe functional abnormalities on the Qualification Echo, unless deemed not clinically relevant by the Investigator and subsequently approved by the Sponsor; ejection fraction (EF, estimated from the Qualification Echo) that is ≤55% (outside normal range), history or clinical manifestations of significant mental illness or significant pulmonary, hematological, renal, hepatic, central nervous, cardiovascular, genitourinary, or gastrointestinal disorders, or diabetes; history of any major surgical procedure within 90 days of Screening/Baseline; body mass index (BMI) >35; sitting systolic blood pressure <90 mmHg or >150 mmHg, diastolic blood pressure <50 mmHg or >95 mmHg, or a pulse rate <45 bpm or >90 bpm; oxygen saturation <92% at rest; and inadequate image quality on the Qualification Echo. Other exclusion criteria include: participation in an investigational drug/device study within 30 days prior to dosing (90 days for UK sites), participation in a previous clinical trial of AI-700, non-seasonal asthma within the past 3 years or recent seasonal asthma requiring prescription medication, frequent (>5/min) premature ventricular or atrial contractions (PVC, PAC), and any ≥2nd AV block, bundle branch block (BBB), or rhythm abnormality.
* Stable cardiac patients in Cohorts A or B who have had any of the following conditions will be excluded from the study: any clinically unstable condition or major surgery within 30 days prior to Screening/Baseline (including but not limited to severe arterial hypertension, pulmonary hypertension, or any increase in pulmonary pressures due to increased pulmonary resistance, hypotension, bradycardia, tachycardia, unstable angina); cerebrovascular accident or transient ischemic attack within 90 days prior to dosing; congestive heart failure graded as New York Heart Association Class 3 or 4 within 90 days prior to dosing; significant left main CAD (≥50% stenosis); moderate to severe chronic obstructive pulmonary disease (COPD) within 6 months prior to dosing; or oxygen saturation <90% at rest; and inadequate image quality on the Qualification Echo. Candidates with clinically significant intra-cardiac shunts or any other cardiovascular structural and/or severe functional abnormalities per the Qualification Echo [including intra cardiac shunts; uncorrected congenital heart disease (i.e., severe valvular disease; large amount of pericardial effusion], EF (as estimated from the Qualification Echo) of <40%; are also not eligible to participate. Subjects who exhibit new or changing ECG abnormalities at any time between Screening and AI-700 dosing will be similarly excluded. Other exclusion criteria include: participation in an investigational drug/device study within 30 days prior to dosing (90 days for UK sites), participation in a previous clinical trial of AI-700, non-seasonal asthma within the past 3 years or recent seasonal asthma requiring prescription medication, organ transplant or end-stage organ failure, and active seizure disorder. Candidates will also be excluded for uncontrolled atrial fibrillation, frequent (>5/min) PVCs or PACs, history of prolonged QT/QTc (>500 msec), use of automatic implantable cardioverter/defibrillator, and any ≥2nd AV block, BBB, or rhythm abnormality that has not been evaluated and treated by a specialist or for which current treatment is not adequately effective to the extent that subject safety is assured.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-11; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Image quality of echocardiographic data collected via several ultrasound imaging platforms
For Cohort B, the duration of MCE following the first 0.04 mL/kg dose of AI-700
Safety of AI-700 administered IV to healthy volunteers and suspected CAD patients

CONTACTS AND LOCATIONS:
Locations (1):
- Acusphere, Inc., Watertown, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.acusphere.com